CLINICAL TRIAL: NCT00135317
Title: A Randomized Open-Label Study of Darbepoetin Alfa Administered Every Three Weeks With or Without Parenteral Iron in Anemic Subjects With Nonmyeloid Malignancies Receiving Chemotherapy
Brief Title: AIM 3: Anemia and Iron Management With Every 3 Week Dosing in Anemic Subjects With Nonmyeloid Malignancies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040156
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Cancer
Keywords: oncology; darbepoetin alfa; Aranesp®; Amgen; Non-myeloid malignancy
MeSH Terms: conditions — Neoplasms | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa

SUMMARY:
The study is designed to assess if the addition of intravenous (IV) iron to 500 mcg every 3 week (Q3W) darbepoetin alfa treatment enhances response as compared to the standard practice (oral iron or no iron administration).

ELIGIBILITY:
Inclusion Criteria: - Subjects with non-myeloid malignancy (chronic myeloid leukemia [CML], acute leukemia [acute myelogenous leukemia (AML) and acute lymphocytic leukemia (ALL)], hairy cell leukemia, Burkitt's lymphoma and lymphoblastic lymphoma are specifically excluded) - Planned to receive at least 8 weeks of cyclic cytotoxic chemotherapy regardless of schedule (chemotherapy may already be ongoing at time of screening) - Hemoglobin concentration less than 11 g/dL within 24 hours before randomization - Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 Exclusion Criteria: - Known (documented in medical records) history of seizure disorder (subjects with a previous history of seizure disorders will be eligible for the study, if they have had no evidence of seizure activity, and have not been taking anti-seizure medication for the previous 5 years) - Known (documented in medical records) history of thromboembolism - Known primary hematologic disorder which could cause anemia other than a non-myeloid malignancy (e.g., sickle cell anemia, thalassemia) - Radiotherapy within 4 weeks before randomization in which the radiation is administered to greater than 25% of the marrow - Unstable or uncontrolled disease/condition, related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension and/or unstable cardiac arrhythmia) - Chronic inflammatory disease that is not stable (e.g., rheumatoid arthritis, Crohn's disease, peptic ulcer, ulcerative disease, etc) - Inadequate renal and/or liver function - Received any red blood cell transfusion within 14 days before randomization or any planned red blood cell transfusion between randomization and study day 1 - Received any erythropoietic therapy within 4 weeks before randomization or any planned erythropoietic therapy between randomization and study day 1 - Known sensitivity to iron administration - Subject of reproductive potential is evidently pregnant (e.g., positive serum HCG test) or is breast feeding - Subject of reproductive potential who is not using adequate contraceptive precautions - Subject has any kind of disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-11

PRIMARY OUTCOMES:
Proportion of subjects achieving a hematopoietic response (hemoglobin [hgb] greater than or equal to 12 g/dL or rise in hgb of greater than 2 g/dL) during the treatment period

SECONDARY OUTCOMES:
Time to hematopoietic response in days
The proportion of subjects with at least one red blood cell (RBC) transfusion from week 5 (day 29) to end of treatment period (EOTP)
Change in hemoglobin from baseline to EOTP
The proportion of subjects achieving a hemoglobin concentration greater than or equal to 11.0 g/dL, in the absence of RBC transfusions in the preceding 28 days, from week 5 to EOTP
The average hgb after achieving a hgb level greater than or equal to 11.0 g/dL
Patient reported outcomes: Change in Functional Assessment of Cancer Therapy (FACT)-Fatigue subscale score from baseline to EOTP
Change in FACT-G Physical Well-being subscale from baseline to EOTP
Change in FACT-G total score from baseline to EOTP
Change in EuroQoL (EQ-5D) thermometer and ED-5D scores from baseline to EOTP

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Bastit L, Vandebroek A, Altintas S, Gaede B, Pinter T, Suto TS, Mossman TW, Smith KE, Vansteenkiste JF. Randomized, multicenter, controlled trial comparing the efficacy and safety of darbepoetin alpha administered every 3 weeks with or without intravenous iron in patients with chemotherapy-induced anemia. J Clin Oncol. 2008 Apr 1;26(10):1611-8. doi: 10.1200/JCO.2006.10.4620. PMID 18375890
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20040156.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf